CLINICAL TRIAL: NCT03906123
Title: The Efficacy of DL-3-n-butylphthalide (DL-NBP) on the Cognitive Function and Vascular Regulation in Patients With Mild Vascular Dementia (VaD) Caused by Subcortical Ischemic Vascular Disease (SIVD)
Brief Title: The Efficacy of DL-NBP in Patients With Mild Subcortical Ischemic Vascular Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Nan Zhang, MD, PhD, Associate Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TianjinMUGH001
Record Dates: First submitted 2019-03-27; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Subcortical Vascular Dementia; Cerebral Small Vessel Diseases
Keywords: DL-3-n-butylphthalide; vascular dementia; cerebral small vessel disease; cognitive function; cerebral blood flow
MeSH Terms: conditions — Dementia, Vascular; Cerebral Small Vessel Diseases | interventions — 3-n-butylphthalide

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBP (Experimental): DL-3-n-butylphthalide (NBP), soft capsule, 200mg Tid, po, for 48 weeks.
  Interventions: Drug: NBP
- Placebos (Placebo Comparator): Placebo, soft capsule, 200mg Tid, po, for 48 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: NBP — NBP soft capsules
  Other Names: DL-3-n-butylphthalide
  Arms: NBP
Drug: Placebos — Soft capsules manufactured to mimic NBP
  Arms: Placebos

SUMMARY:
This is a 48-week, double-blind, randomized, placebo-controlled study. Sixty-four patients are randomly assigned to take NBP (600mg per day) or placebo for 48 weeks, with 32 patients in each treatment group. Anti-dementia treatment-naive patients meet the inclusion/exclusion criteria are enrolled.

Patients are assigned to NBP will take 200mg tid daily. Patients are visited at baseline, as well as 4, 12, 24, 36, 48weeks after baseline. Safety data is recorded until an additional 30 days after the last treatment (48 weeks).

The primary outcomes include cognitive function and activities of daily living (ADL). All subjects are assessed at baseline, 4w, 12w,24w, 36w intermittent visit and 48w endpoint with the Auditory Verbal Learning Test (AVLT), the Brief Visuospatial Memory Test-Revised (BVMT-R), the Symbol Digit Modalities Test (SDMT), the Trail Making Test-A/B (TMT-A/B), the Benton Judgment of Line Orientation (JLO), the verbal fluency test, the Boston Naming Test (BNT), the Controlled Oral Word Association Test (COWAT), the Stroop test, the Mini-Mental State Examination (MMSE), the Montreal Cognitive Assessment (MoCA) and the ADL. The secondary outcomes include the global function and behavioral and psychological symptoms of dementia (BPSD), which are evaluated with the Clinical Dementia Rating (CDR) and the Neuropsychiatric Inventory (NPI), respectively. Independent raters who are blinded to patients' distribution are assigned to assess the participants.

The exploratory outcomes are markers of vascular regulation, including circulating endothelial progenitor cells (EPCs), white matter hyperintensities (WMH) on MRI, cerebral blood flow (CBF) measured with transcranial Doppler (TCD) and arterial spin labeling (ASL) MRI, and parameters of carotid duplex ultrasonic (CDU). In addition, apolipoprotein E (APOE) polymorphism and plasma biomarkers are also detected.

Safety are assessed at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the criteria of major neurocognitive disorder in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
2. Patients aged with 50-80 years, years of education no less than 3, an MMSE range of 15~26, an MoCA < 26, an Hamilton Depression Scale (HAMD) < 17;
3. The MRI (one research dedicated machine 3.0 T) features satisfy subcortical small vessel disease, including (1) multiple (>=3) supratentorial subcortical lacunes (3-20 mm in diameter), with/without white matter hyperintensities (WMH) of any degree; (2) moderate to severe WMH (score>= 2 according to the Fazekas rating scale in either periventricular region or deep white matter) with/without lacunes; (3) one or more strategically located subcortical small infarcts in the deep grey matters;
4. Patients or legal representative should sign the informed consent and have a reliable caregiver.

Exclusion Criteria:

1. Cognitive impairment caused by other central nervous system diseases, such as AD, dementia with Lewy body, frontal-temporal lobe degeneration, etc;
2. Cognitive impairment due to other conditions, such as severe depression, vitamin B 12 deficiency, abnormal thyroid function, etc;
3. Alcoholism, drug abuse or other conditions influenced the evaluation of cognition;
4. Patients unable to undertake MRI assessment.
5. Patients with a history of other severe disease such as epilepsy, myocardial infarction or heart failure will be excluded;
6. Administration of other investigational drugs, psychotropic drugs, drugs with psychiatric side effects, and oral anticoagulants are not allowed

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-11-18 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Auditory Verbal Learning Test (AVLT) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  AVLT is used to evaluate verbal learning and memory ability. Higher score indicates better performance.
Brief Visuospatial Memory Test-Revised (BVMT-R) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  BVMT-R is used to evaluate spatial memory ability. Higher score indicates better performance.
Digital span (DS) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  DS is used to assess attention. Higher score indicates better performance.
Symbol Digit Modalities Test (SDMT) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  SDMT is used to assess information processing speed. Higher score indicates better performance.
Trail Making Test-A (TMT-A) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  TMT-A is used to assess information processing speed. Lower score indicates better performance.
TMT-B at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  TMT-B is used to assess executive function. Lower score indicates better performance.
Stroop test at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  Stroop test is used to assess executive function. Higher score indicates better performance.
Benton Judgment of Line Orientation (JLO) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  JLO is used to assess visuospatial function. Higher score indicates better performance.
Verbal fluency test at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  Verbal fluency test is used to evaluate language function. Higher score indicates better performance.
Boston Naming Test (BNT) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  BNT is used to evaluate language function. Higher score indicates better performance.
Controlled Oral Word Association Test (COWAT) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  COWAT is used to evaluate language function. Higher score indicates better performance.
Mini-Mental State Examination (MMSE) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  MMSE is used to evaluate global cognition. Higher score indicates better performance.
Montreal Cognitive Assessment (MoCA) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  MoCA is used to evaluate global cognition. Higher score indicates better performance.
Activity of daily living (ADL) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  ADL is used to evaluate activities of daily living.

SECONDARY OUTCOMES:
Global function at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  Clinical Dementia Rating (CDR) is used to evaluate global function.
Neuropsychiatric Inventory (NPI) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  NPI is used to evaluate behavioral and psychological symptoms of dementia (BPSD).

OTHER OUTCOMES:
Hamilton Depression Scale (HAMD) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  HAMD is used to evaluate depressive symptoms.
Geriatric Depression Scale (GDS) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  GDS is used to evaluate depressive symptoms.
Regulation of endothelial progenitor cell at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  Circulating endothelial progenitor cell (EPC) is detected with flow cytometry.
Transcranial Doppler (TCD) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  TCD is used to measure cerebral blood flow.
Carotid duplex ultrasonic (CDU) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  CDU is used to evaluate cerebral blood flow and arteriosclerosis.
Arterial spin labeling (ASL) MRI at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  Arterial spin labeling (ASL) is used to measure cerebral blood flow.
White matter hyperintensities (WMH) at endpoint and change from baseline | 48 weeks post-dose and change from baseline
  The extent and volume of WMH are analyzed on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Zhang, MD, PhD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medicial University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.